CLINICAL TRIAL: NCT01019785
Title: Vitamin D During In Vitro Fertilisation (IVF) - A Prospective Randomized Trial
Acronym: Delivery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Pelle G Lindqvist, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Delivery2009
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Pregnancy Complication
Keywords: Pregnancy rate (pos test, live fetus at 12 weeks, baby home); Pregnancy complication (Pregnancy hypertension, SGA, diab); Thrombin generation
MeSH Terms: conditions — Pregnancy Complications; Hypertension, Pregnancy-Induced | interventions — Ergocalciferols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose Vitamin D (Active Comparator)
  Interventions: Dietary Supplement: Ergocalciferol
- Low dose Vitamin D (Sham Comparator)
  Interventions: Dietary Supplement: Ergocalciferol

INTERVENTIONS:
Dietary Supplement: Ergocalciferol — 100 000 U drops is given once
  Other Names: Made by the Swedish APOTEKET
  Arms: High dose Vitamin D
Dietary Supplement: Ergocalciferol — 500 U drops given once
  Arms: Low dose Vitamin D

SUMMARY:
During IVF treatment women will be randomized into supplementation with a high or a low dose of Vitamin D Main outcome Laboratory pregnancy, live pregnancy at 12 weeks, Baby take home rate, OHSS Secondary outcome: 1. Pregnancy complications (pregnancy hypertension, SGA, Diabetes) 2.Thrombin generation

ELIGIBILITY:
Inclusion Criteria:

* All women initiating IVF treatment

Exclusion Criteria:

* Women that have entered the study before

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Laboratory pregnancy, live pregnancy at 12 weeks, take home baby rate | 4 weeks to 9 month

SECONDARY OUTCOMES:
Pregnancy complications (pregnancy hypertension, SGA, diabetes) | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- IVF Unit Karolinska University Hospital, Huddinge, Huddinge, Sweden

REFERENCES:
- [Background] Epstein E, Lindqvist PG, Geppert B, Olsson H. A population-based cohort study on sun habits and endometrial cancer. Br J Cancer. 2009 Aug 4;101(3):537-40. doi: 10.1038/sj.bjc.6605149. Epub 2009 Jun 23. PMID 19550419
- [Background] Lindqvist PG, Epstein E, Olsson H. Does an active sun exposure habit lower the risk of venous thrombotic events? A D-lightful hypothesis. J Thromb Haemost. 2009 Apr;7(4):605-10. doi: 10.1111/j.1538-7836.2009.03312.x. PMID 19335448
- [Derived] Showell MG, Mackenzie-Proctor R, Jordan V, Hart RJ. Antioxidants for female subfertility. Cochrane Database Syst Rev. 2020 Aug 27;8(8):CD007807. doi: 10.1002/14651858.CD007807.pub4. PMID 32851663